CLINICAL TRIAL: NCT00006093
Title: A Phase I/II Trial of EMD 121974 for Treatment of Patients With Recurrent Anaplastic Gliomas
Brief Title: EMD 121974 in Treating Patients With Progressive or Recurrent Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068098; NABTT-9911; JHOC-NABTT-9911
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2003-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma | interventions — Cilengitide

INTERVENTIONS:
Drug: cilengitide

SUMMARY:
RATIONALE: EMD 121974 may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: Phase I/II trial to study the effectiveness of EMD 121974 in treating patients who have progressive or recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of EMD 121974 in patients with progressive or recurrent malignant glioma.
* Determine the 6-month progression-free survival, clinical response rate, duration of progression-free survival, and overall survival in patients treated with this drug.
* Determine the effects of this drug on tumor perfusion, measured with magnetic resonance perfusion scan, and markers for angiogenesis in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive EMD 121974 IV over 1 hour twice weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 6-12 patients receive escalating doses of EMD 121974 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which more than 2 of 6 or 4 of 12 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at the MTD.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A minimum of 6 patients will be accrued for phase I of this study within 2-3 months. A total of 23-38 patients will be accrued for phase II of this study within 5-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma that is progressive or recurrent after radiotherapy and/or chemotherapy

  * Eligible subtypes:

    * Anaplastic astrocytoma
    * Anaplastic oligodendroglioma
    * Glioblastoma multiforme
  * Prior low-grade glioma that has progressed to a high-grade glioma (by biopsy) after radiotherapy and/or chemotherapy allowed
* Measurable disease by volumetric and magnetic resonance perfusion scan
* Prior biopsy or resection of recurrent brain tumor allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* Transaminases no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No advanced coronary artery disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious concurrent infection or medical illness that would preclude study
* No other malignancy within the past 5 years except curatively treated carcinoma in situ or basal cell skin cancer
* No history of wound healing disorders
* No peptic ulcer disease within the past year
* Mini mental score of at least 15
* Willing and able to undergo MRI

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent filgrastim (G-CSF)

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No more than 2 prior chemotherapy regimens

Endocrine therapy:

* Prior corticosteroids allowed if on stable dose for at least 5 days prior to study
* Concurrent corticosteroids (e.g., dexamethasone) allowed as clinically needed

Radiotherapy:

* See Disease Characteristics
* At least 3 months since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics
* At least 1 week since prior surgery and recovered
* No concurrent elective surgery or dental extractions

Other:

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis B. Nabors, MD, Study Chair — University of Alabama at Birmingham
Locations (10):
- United States (10):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Result] Nabors LB, Mikkelsen T, Rosenfeld SS, Hochberg F, Akella NS, Fisher JD, Cloud GA, Zhang Y, Carson K, Wittemer SM, Colevas AD, Grossman SA. Phase I and correlative biology study of cilengitide in patients with recurrent malignant glioma. J Clin Oncol. 2007 May 1;25(13):1651-7. doi: 10.1200/JCO.2006.06.6514. PMID 17470857
- [Result] Nabors LB, Rosenfeld SS, Mikkelsen T, et al.: NABTT 9911: a phase I trial of EMD 121974 for treatment of patients with recurrent malignant gliomas. [Abstract] Neuro-Oncology 6 (4): TA-39, 379, 2004.